CLINICAL TRIAL: NCT04729751
Title: Open-Label, Phase 2 Study to Evaluate the Safety and Tolerability of Maralixibat in the Treatment of Infants With Cholestatic Liver Diseases Including Progressive Familial Intrahepatic Cholestasis and Alagille Syndrome
Brief Title: A Study to Evaluate the Safety and Tolerability of Maralixibat in Infant Participants With Cholestatic Liver Diseases Including Progressive Familial Intrahepatic Cholestasis (PFIC) and Alagille Syndrome (ALGS).
Acronym: RISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRX-801; 2020-004628-40 (EudraCT Number)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Progressive Familial Intrahepatic Cholestasis; Alagille Syndrome; Cholestatic Liver Disease
Keywords: PFIC; ALGS; Maralixibat; Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases; Pediatric
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Alagille Syndrome; Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases | interventions — maralixibat

STUDY DESIGN:
Intervention Model Description: Single group with 2 cohorts - ≥ 6 participants each from ALGS and PFIC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Maralixibat (Experimental): Participants will receive up to 600 μg/kg twice daily (PFIC) or up to 400 μg/kg once daily (ALGS) over 13 weeks in the core study and for the duration of the Long Term Extension (LTE) where applicable.
  Interventions: Drug: Maralixibat

INTERVENTIONS:
Drug: Maralixibat — Maralixibat chloride provided in the form of an oral solution (i.e., 5, 10, 15, and 20 mg/mL)
  * 400 μg/kg maralixibat chloride is equivalent to 380 µg/kg maralixibat free base
  * 600 μg/kg maralixibat chloride is equivalent to 570 µg/kg maralixibat free base
  Other Names: Formerly LUM001 and SHP625

SUMMARY:
This study is designed to assess whether the investigational drug maralixibat, is safe and well tolerated in children <12 months of age with Alagille Syndrome [ALGS] or Progressive Familial Intrahepatic Cholestasis [PFIC].

DETAILED DESCRIPTION:
This is an open label study where all participants will receive maralixibat treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight of ≥2.5 kg
2. <12 months of age at the baseline visit (ROW). >31 days and <12 months of age at the baseline visit (US).
3. Gestational age ≥36 weeks at birth. For children born with gestational age between 32 and 36 weeks, a postmenstrual age of ≥36 weeks is required.
4. Diagnosis of PFIC or ALGS

Exclusion criteria:

1. Predicted complete absence of bile salt excretion pump (BSEP) function
2. History of surgical disruption of the enterohepatic circulation
3. History of liver transplant or imminent need for liver transplant
4. Decompensated cirrhosis
5. Presence of any other disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, including bile salt metabolism in the intestine (e.g., inflammatory bowel disease), per investigator discretion
6. Presence of other significant liver disease or any other conditions or abnormalities which, in the opinion of the investigator or medical monitor, may compromise the safety of the participant or interfere with the participant's participation in or completion of the study

Ages: 0 Days to 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events [TEAEs] | From Baseline through to Week 13

SECONDARY OUTCOMES:
Change in fasting serum bile acid (sBA) levels | From Baseline through to Week 13
To evaluate the effect on liver enzymes (ALT, AST) and bilirubin | From Baseline through to Week 13
To evaluate the effect on LSVs | From Baseline through to Week 13
To assess the plasma level of maralixibat in infant participants | At Baseline, Week 6, Week 10, Week 13 or Early Termination Visit

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - Children Hospital LA, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Ochsner Hospital for Children, New Orleans, Louisiana
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Sociedade Beneficente de Senhoras - Hospital Sírio-Libanês, São Paulo, Brazil
- France (2):
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hopital Necker, Paris
- Consultorio de Joshue David Covarrubias Esquer, Zapopan, Mexico
- Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Poland
- King's College Hospital, London, United Kingdom

REFERENCES:
- See also: Genetics Home Reference - PFIC — https://medlineplus.gov/genetics/condition/progressive-familial-intrahepatic-cholestasis/
- See also: Mirum Pharmaceuticals homepage — https://mirumpharma.com
- See also: Genetics Home Reference - ALGS — https://medlineplus.gov/genetics/condition/alagille-syndrome/
- See also: US FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks